CLINICAL TRIAL: NCT04166721
Title: A Multicenter Phase II Non-randomised Trial Assessing the Efficacy of DKN-01 Plus Atezolizumab in Patients With Advanced Mismatch Repair Proficient Oesophagogastric Cancer
Brief Title: WaKING: Wnt and checKpoint INhibition in Gastric Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCR4976
Record Dates: First submitted 2019-11-12; First posted 2019-11-18 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Esophageal Cancer; Metastatic Gastric Cancer
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms | interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DKN-01 and atezolizumab (Experimental): DKN-01 is an intravenous medication which will be given at a variable dose during the Phase IIA safety run in phase of the trial (150mg, 300mg or 600mg IV q14d).
  During the Phase IIB efficacy phase of the trial patients will be treated with DKN-01 at the safe and tolerated combination dose identified during the Phase IIA safety run in phase.
  Atezolizumab is a monoclonal antibody which is given via an intravenous infusion at a dose of 840mg on the first day of a two week cycle. (Day 1 q 14d) from cycle 2 onwards.
  In the first cycle of treatment, patients will be treated with only DKN-01, and following this they will be treated with both DKN-01 and atezolizumab
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: Atezolizumab — Immunotherapy
  Other Names: DKN-01

SUMMARY:
This is a multicentre open-label non-randomised, Single Stage Ahern Design (with a 3+3 design for the safety run-in) phase II clinical trial of DKN-01 plus atezolizumab in patients with advanced unresectable or metastatic OGA who have progressed following chemotherapy.

DETAILED DESCRIPTION:
A multi-centre phase II open label non-randomised trial of DKN-01 plus atezolizumab in patients with advanced inoperable or metastatic mismatch repair proficient gastroesophageal cancer (GC) who have progressed following chemotherapy. This trial is designed to evaluate the safety and efficacy of administering DKN-01, a DKK1 inhibitor plus atezolizumab, an anti-PD-L1 monoclonal antibody in this patient cohort. This trial is in 2 stages: the first stage (Phase IIA, 3+3 safety run-in) will establish a safe and tolerated dose of DKN-01 in combination with atezolizumab and the second stage (Phase IIB, Single Stage A'hern design for efficacy/ anti-tumour activity) will assess the efficacy of this combination therapy in achieving tumour response according to RECIST 1.1 criteria (additional iRECIST criteria will be used in a sensitivity analysis).

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form
2. Male or female patients age ≥18 years at time of signing Informed Consent Form
3. Ability to comply with the study protocol, in the investigator's judgment
4. Histologically or cytologically confirmed advanced or metastatic gastroesophageal adenocarcinoma. Patients with HER2 positive cancer are permitted after having received HER2 targeted therapy in first line as per Standard of Care
5. Disease progression during or following treatment with one or two lines of treatment for advanced disease, one of which must have been a platinum and fluoropyrimidine combination.
6. Measurable, or non-measurable but evaluable, disease per RECIST v1.1
7. Evidence of tumor mismatch repair proficiency and/or MSI stability through testing of a representative tumor tissue specimen using immunohistochemistry for MMR proteins or MSI testing. Local testing or historical results of archival tumour tissue is satisfactory for trial entry.
8. ECOG 0-1
9. Life expectancy ≥ 3 months as per physician judgment
10. Adequate hematologic and end-organ function, defined by the following laboratory test results:

    a. ANC ≥ 1.5 x 109/L without granulocyte colony-stimulating factor support b. Lymphocyte count ≥ 0.5 x 109/L c. Platelet count ≥ 100 x 109/L without transfusion d. Hemoglobin ≥ 90 g/L (9 g/dL) (patients may be transfused to meet this criterion) e. AST, ALT, and alkaline phosphatase (ALP) ≤ 2.5 x upper limit of normal (ULN), with the following exceptions: i. Patients with documented liver metastases: AST and ALT ≤ 5 x ULN ii. Patients with documented liver or bone metastases: ALP ≤ 5 x ULN f. Serum bilirubin ≤ 1.5 x ULN with the following exception: i. Patients with known Gilbert disease: serum bilirubin level ≤ 3 x ULN g. Serum creatinine ≤ 1.5 x ULN or Creatinine clearance (CrCl) ≥ 50 mL/min (calculated using the Cockcroft-Gault formula)} h. Serum albumin ≥ 25 g/L (2.5 g/dL) i. For patients not receiving therapeutic anticoagulation: INR or aPTT ≤ 1.5 x ULN j. For patients receiving therapeutic anticoagulation: stable anticoagulant regimen k. Negative hepatitis B surface antigen (HBsAg) test at screening l. Negative total hepatitis B core antibody (HBcAb) test at screening, or positive total HBcAb test followed by quantitative hepatitis B virus (HBV) DNA < 500 IU/mL at screening m. The HBV DNA test will be performed only for patients who have a positive total HBcAb test.

    n. Negative hepatitis C virus (HCV) antibody test at screening, or positive HCV antibody test followed by a negative HCV RNA test at screening o. The HCV RNA test will be performed only for patients who have a positive HCV antibody test.
11. Tumour is amenable to safe repeated biopsies and patient agrees to undergo biopsies for translational endpoints.
12. In patients who are receiving anticoagulation, stopping anticoagulation for biopsies must be deemed safe by the treating team.
13. Patients on oral anticoagulation are required to change to low molecular weight heparin prior to study entry to be eligible.
14. Willingness and ability to comply with the protocol for the duration of the study including scheduled visits, examinations, investigations and treatment plans
15. Pregnancy must be excluded with a negative serum pregnancy test, within 7 days before initiation of therapy, if the risk of conception exists.

Exclusion Criteria:

1. Any contraindication or known hypersensitivity reaction to any of the study drugs
2. Persisting toxicity relating to prior therapy of >grade 1 CTCAE version 5.0 except alopecia of any grade and neuropathy ≤ grade 2, or other grade ≤2 not constituting a safety risk based on investigators judgement
3. Any prior treatment with immunotherapy including anti-PD-1or PD-L1 therapy
4. known active or untreated CNS metastases are excluded. Patients with treated and asymptomatic CNS metastases are eligible, if they meet all of the following:

   1. Evaluable or measurable disease outside the CNS
   2. No metastases to midbrain, pons, medulla, or within 10 mm of the optic nerves and chiasm
   3. No history or evidence of intracranial haemorrhage or spinal cord haemorrhage
   4. No evidence of clinically significant vasogenic oedema
   5. Not on corticosteroids for ≥ 2 weeks; anti-convulsants at a stable dose are allowed
   6. No evidence of clinical and radiographic disease progression in the CNS ≥ 3 weeks after radiotherapy or surgery
5. Known severe hypersensitivity reactions to monoclonal antibodies (Grade ≥ 3 NCI CTCAE v 5.0), any history of anaphylaxis
6. Any Immunodeficiency disorder
7. Patients with another active malignancy or a prior malignancy within the past 5 years are excluded, except patients with completely resected cutaneous melanoma (early stage), basal cell carcinoma, cutaneous squamous cell carcinoma, cervical carcinoma in-situ, breast carcinoma in-situ, and localized prostate cancer are eligible
8. History of autoimmune disease except for the following:

   1. Patients with autoimmune hypothyroidism on a stable dose of thyroid replacement hormone are eligible
   2. Patients with controlled type 1 diabetes mellitus on a stable dose of insulin regimen are eligible
   3. Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g. patients with psoriatic arthritis) are permitted provided that they meet the following conditions:

      * Patients with psoriasis must have a baseline ophthalmologic exam to rule out ocular manifestations
      * Rash must cover less than 10% of body surface area
      * Disease is well controlled at baseline and only requiring low-potency topical steroids (e.g., hydrocortisone 2.5%, hydrocortisone butyrate 0.1%, flucinolone 0.01%, desonide 0.05%, aclometasone dipropionate 0.05%)
      * No acute exacerbations of underlying condition within the last 12 months (not requiring PUVA [psoralen plus ultraviolet A radiation], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral steroids)
9. History of idiopathic pulmonary fibrosis, organizing pneumonia, bronchiolitis obliterans, drug-induced pneumonitis, or idiopathic pneumonitis Patients with radiation pneumonitis within the radiation field are eligible

12. Prior organ transplantation, including allogeneic transplant 13. Significant infection requiring systemic therapy 14. Known positive tests for human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome 15. History of inflammatory bowel disease 16. History of stroke, reversible ischemic neurological defect, or transient ischemic attack within 6 months prior to Day 1

17. Proteinuria >grade 1 (≥ ULN - ≤1.0g/24hr) 18. Serum albumin < 2.5 g/dL 19. Administration of a live, attenuated vaccine within 4 weeks before randomization or anticipation of a live attenuated vaccine will be required during the study 20. Treatment with systemic immunostimulatory agents (including but not limited to interferons, IL-2) within 4 weeks or 5 half-lives of the drug, whichever is shorter, prior to Cycle 1 Day 1 21. Treatment with systemic immunosuppressive medications (including but not limited to prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumour necrosis factor [TNF] agents) within 2 weeks prior to Cycle 1 Day 1 22. Cardiovascular diseases as follows:

1. Unstable angina, new onset angina within last 3 months, myocardial infarction within last 6 months and current congestive heart failure New York Heart Association Class II or higher.
2. Left ventricular ejection fraction (LVEF) below institutional lower limit of normal or below 50%, whichever is lower.
3. Poorly controlled hypertension, defined as a blood pressure consistently above 150/90 mmHg despite optimal medical management.

   23. Current signs or symptoms of any other severe progressive or uncontrolled hepatic, hematologic, gastrointestinal, endocrine, respiratory or cardiac disease, which in the opinion of the investigator, might impair the subject's tolerance of trial treatment or procedures.

   24. Major surgery, major trauma or open biopsy within 28 days prior to registration (not including staging laparoscopy) 25. Evidence of bleeding diathesis or coagulopathy 26. Active non-healing wound, ulcer or bone fracture requiring therapy 27. Current lactation. Patients who agree to stop breastfeeding may be eligible.

   28. Other severe acute or chronic medical conditions or psychiatric conditions including recent (within the past year) or active suicidal ideation or behaviour; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

   29. Uncontrolled tumour-related pain. Patients requiring narcotic pain medication must be on a stable regimen at study entry. Symptomatic lesions (e.g., bone metastases or metastases causing nerve impingement) amenable to palliative radiotherapy should be treated prior to start of study treatment.

   30. Uncontrolled pleural effusion, pericardial effusion or ascites requiring repeated drainage more than once every 28 days. Indwelling drainage catheters (e.g., PleurX®) are allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2020-02-11 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety run-in phase: To recommend a safe and tolerable dose of combination DKN-01 and atezolizumab for use in the main (Phase IIB efficacy) phase of this trial. | The DLT period is 28 days from the start of the combination of DKN-01 and atezolizumab for any given patient (i.e. from C2 D1)
  Progression through dose levels will be determined by the occurence of dose limiting toxicities in the study population
Main phase IIB (efficacy) phase: Best objective response rate (ORR) using RECIST 1.1 criteria | 24 months
  ORR will be defined in the mITT population as the proportion of patients who have achieved CR or PR (as assessed according to RECIST 1.1 criteria) as their best overall response during treatment. The rate will be presented as a proportion with an exact 95% confidence interval.

SECONDARY OUTCOMES:
The safety of DKN-01 plus atezolizumab will be assessed in the Safety Population (SFP) according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0 | Up to 135 days after the last dose
Progression free survival (PFS) according to RECIST 1.1 | Up to 24 months
  PFS will be estimated in the mITT population using the Kaplan Meier method and presenting median survival with 95% confidence intervals. 6 month and 1 year PFS will also be reported. PFS will be defined as time from first drug administration (C1D1) to clinical/radiological progression or death from any cause.
Overall survival | Up to 24 months
  OS will be estimated in the mITT population using the Kaplan Meier method and presenting median survival with 95% confidence intervals. 6 month and 1 year OS will also be reported. PFS will be defined as time from first drug administration (C1D1) to clinical/radiological progression or death from any cause and OS will be defined time from first drug administration (C1D1) to date of death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR